CLINICAL TRIAL: NCT03196466
Title: Population Pharmacokinetics of Antiepileptic in Pediatrics
Acronym: EPIPOP
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: NI17009HLJ
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Epilepsy
Keywords: antiepileptics; pharmacokinetics; children; genetic polymorphisms
MeSH Terms: conditions — Epilepsy | interventions — Valproic Acid; Carbamazepine; Phenobarbital; Phenytoin; Levetiracetam; Lamotrigine; Topiramate; Oxcarbazepine; stiripentol; Clobazam; Felbamate; Lacosamide; rufinamide; Gabapentin; sulthiame; Tiagabine; Vigabatrin; methsuximide; Primidone; perampanel; Ethosuximide; Zonisamide; Cannabidiol; Polymorphism, Genetic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- antiepileptics titration: Titration of valproic acid, carbamazepine, phenobarbital, phenytoin, levetiracetam, lamotrigine, topiramate, oxcarbazepine, stiripentol, clobazam, brivaracétam, felbamate, lacosamide, rufinamide, gabapentine, pregabaline, sultiame, tiagabine, vigabatrine, mesuximide, primidone, perampanel, ethosuximide, zonisamide and cannabidiol
  Interventions: Biological: Valproic acid; Biological: carbamazepine; Biological: phenobarbital; Biological: phenytoin; Biological: levetiracetam; Biological: lamotrigine; Biological: topiramate; Biological: oxcarbazepine; Biological: stiripentol; Biological: clobazam; Biological: brivaracétam; Biological: felbamate; Biological: lacosamide; Biological: rufinamide; Biological: gabapentine; Biological: pregabaline; Biological: sultiame; Biological: tiagabine; Biological: vigabatrine; Biological: mesuximide; Biological: primidone; Biological: perampanel; Biological: ethosuximide; Biological: zonisamide; Biological: cannabidiol
- antiepileptics titration and available blood samples: Titration of valproic acid, carbamazepine, phenobarbital, phenytoin, levetiracetam, lamotrigine, topiramate, oxcarbazepine, stiripentol, clobazam, brivaracétam, felbamate, lacosamide, rufinamide, gabapentine, pregabaline, sultiame, tiagabine, vigabatrine, mesuximide, primidone, perampanel, ethosuximide, zonisamide and cannabidiol
  Interventions: Biological: Valproic acid; Biological: carbamazepine; Biological: phenobarbital; Biological: phenytoin; Biological: levetiracetam; Biological: lamotrigine; Biological: topiramate; Biological: oxcarbazepine; Biological: stiripentol; Biological: clobazam; Biological: brivaracétam; Biological: felbamate; Biological: lacosamide; Biological: rufinamide; Biological: gabapentine; Biological: pregabaline; Biological: sultiame; Biological: tiagabine; Biological: vigabatrine; Biological: mesuximide; Biological: primidone; Biological: perampanel; Biological: ethosuximide; Biological: zonisamide; Biological: cannabidiol; Other: genetic polymorphisms

INTERVENTIONS:
Biological: Valproic acid — titration
Biological: carbamazepine — titration
Biological: phenobarbital — titration
Biological: phenytoin — titration
Biological: levetiracetam — titration
Biological: lamotrigine — titration
Biological: topiramate — titration
Biological: oxcarbazepine — titration
Biological: stiripentol — titration
Biological: clobazam — titration
Biological: brivaracétam — titration
Biological: felbamate — titration
Biological: lacosamide — titration
Biological: rufinamide — titration
Biological: gabapentine — titration
Biological: pregabaline — titration
Biological: sultiame — titration
Biological: tiagabine — titration
Biological: vigabatrine — titration
Biological: mesuximide — titration
Biological: primidone — titration
Biological: perampanel — titration
Biological: ethosuximide — titration
Biological: zonisamide — titration
Biological: cannabidiol — titration
Other: genetic polymorphisms — genetic polymorphisms
  Groups: antiepileptics titration and available blood samples

SUMMARY:
The purpose of this study is to develop population pharmacokinetic models for antiepileptic drugs in a pediatric population.

The interest of these models is multiple:

* describe the pharmacokinetics of these molecules in children and explain the inter-individual variability of concentrations through covariates such as weight, age, co-treatments, genetic polymorphisms and renal function;
* estimate maximum, minimum and exposure concentrations from the individual pharmacokinetic parameters for each patient;
* propose adaptations of doses for certain classes of children (according to age, weight etc.) and individualize the doses.

DETAILED DESCRIPTION:
Epilepsy affects about 1% of the population, with a peak incidence in childhood, and persistent seizures on antiepileptic therapy in approximately 30% of patients. Over the past two decades, many antiepileptic molecules have emerged, raising the question of their optimal use, especially in pediatrics, where pharmacokinetics and pharmacodynamics are different from adults and largely influenced by age and development.

The pharmacokinetics of antiepileptics have been little studied in pediatric populations. In children, it is important to know if a maturational effect (of age) has to be taken into account in addition to the physiological effect (of the weight) to adapt the doses. Moreover, these molecules are often used in combination and lot of enzyme interactions make their use delicate. All of these factors explain the existence of significant inter-individual variability in the pediatric population.

The implication of the demographic and medicinal factors mentioned above, as well as the balance of efficacy / undesirable effects, justify the interest of a pharmacological monitoring of these drugs in a pediatric population. The use of population pharmacokinetics is particularly interesting in children because it requires only a small number of samples per patient and can be used to describe the predominant inter-individual variability in this population.

The main goal is to develop population pharmacokinetic models for the following antiepileptic drugs in children: valproic acid, carbamazepine, phenobarbital, phenytoin, levetiracetam, lamotrigine, topiramate, oxcarbazepine, stiripentol, clobazam, brivaracétam, felbamate, lacosamide, rufinamide, gabapentine, pregabaline, sultiame, tiagabine, vigabatrine, mesuximide, primidone, perampanel, ethosuximide, zonisamide and cannabidiol. The interest of these models is multiple:

* describe the pharmacokinetics of these molecules in children and explain the interindividual variability of concentrations through covariates such as weight, age, co-treatments, genetic polymorphisms and renal function;
* estimate maximum, minimum and exposure concentrations from the individual pharmacokinetic parameters for each patient;
* propose adaptations of doses for certain classes of children (according to age, weight etc.) and individualize the doses.

The secondary objectives of this work are:

* Build models jointly with several antiepileptic drugs, accounting for the strength of interactions between them during multiple therapies.
* Link antiepileptic concentrations to the effects of treatment (reduction or cessation of seizures): pharmacokinetic-pharmacodynamic study with concentration / efficacy and concentration / toxicity relationships.
* The evaluation of preexisting models in the literature and the comparison of the data with the results of these models (external validation).

Pharmaco-statistical analysis will be carried out on the retrospective data of patients treated with one or more antiepileptic molecule (s) and whose blood dosage of the drug(s) as part of their therapeutic follow-up is available. The study of genetic polymorphisms will be carried out from available blood samples, collected and stored as part of therapeutic follow-up of patients.

ELIGIBILITY:
Inclusion Criteria:

* Children from 0 to 18 years of age with epilepsy;
* Treatment with one or more antiepileptic drug (s) studied (valproic acid, carbamazepine, phenobarbital, phenytoin, levetiracetam, lamotrigine, topiramate, oxcarbazepine, stiripentol, clobazam, brivaracétam, felbamate, lacosamide, rufinamide, gabapentine, pregabaline, sultiame, tiagabine, vigabatrine, mesuximide, primidone, perampanel, ethosuximide, zonisamide and cannabidiol);
* Blood dosage of the drug (s) as part of their therapeutic follow-up in the Pharmacology laboratory of the Cochin hospital between 2007 and 2019

Exclusion Criteria:

* patient with missing data on time of last drug taking, time of collection, co-treatments and / or dose administered;
* patient with doubt about compliance

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Minor patient treated by one or more antiepileptics and for which a blood test has been performed
Sampling Method: Non-Probability Sample
Enrollment: 753 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Volume of distribution | through study completion, an average of 5 years
Absorption constant | through study completion, an average of 5 years
Clearance | through study completion, an average of 5 years

SECONDARY OUTCOMES:
Composite measure of the inter-individual variability | through study completion, an average of 5 years
  Covariates of inter-individual variability : age, weight, co-treatments, genetic polymorphisms and renal function

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc TRELUYER, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- AP-HP Cochin, Paris, France

IPD SHARING:
Plan to Share IPD: No